CLINICAL TRIAL: NCT01210534
Title: Physiological Brain Atlas Development
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: 2010H0036
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease; Dystonia; Tremors; Obsessive Compulsive Disorder; Depression
MeSH Terms: conditions — Parkinson Disease; Dystonia; Tremor; Obsessive-Compulsive Disorder; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — No intervention
  Other Names: Single Arm Group

SUMMARY:
Enrollment of candidates undergoing a deep brain stimulator (DBS) implant.

DETAILED DESCRIPTION:
The study proposes the enrollment of candidates undergoing a deep brain stimulator (DBS) implant. Data will be collected before, during and after surgery and will be electronically entered into the Atlas database where it will be stored indefinitely.

The purpose of the study is to create an Atlas to store physiological information utilizing non-rigid MRI normalization algorithms. In addition to collating and analyzing the physiological atlas in a statistical manner that allows the surgeon to predict optimal targeting locations for DBS implants based on multiple physiological variables, including pre-operative severity of disease, intraoperative neurophysiological observations, and post-operative response to DBS stimulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Any patient between the age of 7-90
* Patients who have undergone deep brain stimulation (DBS) surgery as standard of care at The Ohio State University

Exclusion Criteria:

* None

Ages: 7 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are undergoing DBS implantation surgery at the Ohio State University.
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2010-08; Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
optimal DBS target location | intra-operative identification
  To create an atlas that will allow physiological information to be assigned to anatomical locations in MRI space, utilizing non-rigid MRI normalization algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Vibhor Krishna, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio Sate University, Columbus, Ohio, United States